CLINICAL TRIAL: NCT06170255
Title: Depression Treatment and Risk for Cardiovascular Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Matthew Whited, Associate Professor of Psychology, East Carolina University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5K23HL109620 (NIH)
Record Dates: First submitted 2023-11-17; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Depression treatment (Experimental): Participants receive behavioral therapy for depression
  Interventions: Behavioral: Behavioral Activation (BA)

INTERVENTIONS:
Behavioral: Behavioral Activation (BA) — Behavioral activation involves an exploration of the patient's individualized values and follows with goal setting to improve depression symptoms.

SUMMARY:
This study was designed to determine the feasibility of a Randomized Controlled Trial (RCT) that involved treating depression among participants with an elevated risk for cardiovascular disease. It is expected that treating depression through non-pharmacological means will impact heart rate variability, a proximal measure of CVD risk.

ELIGIBILITY:
Inclusion Criteria:

Males and females age 21-75

Meet diagnostic criteria for major depressive disorder

Framingham risk score indicating a greater than negligible 10-year risk (3% or greater) for cardiovascular disease.

Levels of depressive symptoms of at least moderate level (beck depression inventory II score > 19 of 63 possible points; or a Hamilton depression rating scale > 12 of 50 possible points)

Exclusion Criteria:

A verbal expression of current, significant, suicidal ideation; a score of > 15 on the beck scale for suicidal ideation

Score of >1 on any single item of the Beck Scale for Suicidal Ideation

Score of > 1 on the item assessing suicidal ideation on the beck depression inventory II.

Psychiatric diagnoses that could potentially interfere with depression treatment (current post traumatic stress disorder, bipolar I disorder, obsessive-compulsive disorder, bulimia or anorexia nervosa, schizophrenia, and panic disorder)

Current use of an antidepressant medication

Currently in psychotherapy.

Current use of a beta blocker, anxiolytic (benzodiazepine), antipsychotic agent

Diagnosis of CVD.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-03-06 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Feasibility | 2 years. Throughout the course of the study (number recruited/screened, number enrolled, number completing the study)
  Feasibility of the study including recruitment, enrollment, and retention rates

SECONDARY OUTCOMES:
Heart Rate Variability (HRV) | 12 weeks
  Change in HRV from enrollment to post-treatment